CLINICAL TRIAL: NCT00004658
Title: Phase II Study of Ribose, Uridine, and Thymidine for a Complex Syndrome Involving Excessive 5'-Nucleotidase Activity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, San Diego (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11828; UCSD-782
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: 5'-Nucleotidase Syndrome
Keywords: 5'-nucleotidase syndrome; inborn errors of metabolism; rare disease
MeSH Terms: conditions — 5-Nucleotidase syndrome; Metabolism, Inborn Errors; Rare Diseases | interventions — Ribose; Thymidine; Uridine

INTERVENTIONS:
Drug: ribose
Drug: thymidine
Drug: uridine

SUMMARY:
OBJECTIVES: I. Evaluate the efficacy of oral ribose in patients with a complex 5'-nucleotidase syndrome who have not received uridine (UR) and thymidine (TDR).

II. Evaluate the efficacy of UR/oral ribose and UR/TDR. III. Evaluate the efficacy of oral ribose given in combination with UR/TDR.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Newly identified patients receive ribose daily for 8 weeks. Patients who improve continue therapy. If improvement then reaches a plateau, uridine (UR) and thymidine (TDR) are added to the regimen.

Patients who receive no benefit after 8 weeks of ribose are treated with UR/TDR. Patients who improve after 8 weeks of this combination continue therapy.

Ribose is added to the treatment regimen for patients on UR/TDR at entry. At maximal improvement, TDR and UR are sequentially tapered.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Complex syndrome with excessive skin fibroblast 5'-nucleotidase activity characterized by: Recurrent infection Seizure disorder Speech impairment Attention deficit and behavior problems --Prior/Concurrent Therapy-- Concurrent uridine and thymidine therapy allowed --Patient Characteristics-- Other: No pregnant women

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1995-03

CONTACTS AND LOCATIONS:
Overall Officials: Alice L. Yu, Study Chair — University of California, San Diego